CLINICAL TRIAL: NCT06514729
Title: The Effects of Different Ventilation Modes on Patients With Plasma Inflammatory Factor and Respiratory Function in Patients With Pulmonary Lobe Resection
Brief Title: The Effects of Different Ventilation Modes on Patients With Pulmonary Lobe Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mao Enting (Other)
Responsible Party: Sponsor-Investigator, Mao Enting, Anesthesiology resident,Affiliate Hospital of Zunyi Medical University, Zunyi Medical College
Organization: Zunyi Medical College (Other)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: KLL-2023-216
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Lung Injury; Lung Inflammation
MeSH Terms: conditions — Lung Injury; Pneumonia

STUDY DESIGN:
Intervention Model Description: This study was divided into 3 groups, one groups was ventilation side volume control ventilation+continuous positive pressure ventilation on the non ventilation side, the other groups was ventilation side volume control ventilation+continuous positive pressure ventilation on the non ventilation side; the other groups was ventilation side pressure regulated volume control ventilation+continuous positive pressure ventilation on the non ventilation side.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The researchers in this study enrolled suitable patients using a random number table method before surgery, and then performed different intraoperative single lung ventilation modes according to the grouping after unblinding the patients upon entering the room. The postoperative follow-up personnel or data analysts are unaware of the grouping status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group VCV+CPAP (Experimental): Ventilation side volume control ventilation+continuous positive pressure ventilation on the non ventilation side
  Interventions: Procedure: Adopting different ventilation modes during the operation
- Group PCV+CPAP (Experimental): Ventilation side pressure control ventilation+continuous positive pressure ventilation on the non ventilation side
  Interventions: Procedure: Adopting different ventilation modes during the operation
- Group PRVC+CPAP (Experimental): Ventilation side pressure regulated volume control ventilation+continuous positive pressure ventilation on the non ventilation side
  Interventions: Procedure: Adopting different ventilation modes during the operation

INTERVENTIONS:
Procedure: Adopting different ventilation modes during the operation — The ventilation side adopts different ventilation modes combined with continuous positive pressure ventilation on the surgical side.

SUMMARY:
The objective of this study was to discuss the effects of different ventilation modes on patients with plasma inflammatory factor and respiratory function in patients with pulmonary removal.

DETAILED DESCRIPTION:
Patients who meet the inclusion criteria will be numbered in the order of admission, and a dedicated person will prepare codes and opaque envelopes for random allocation. This study was divided into 3 groups, one groups was ventilation side volume control ventilation+continuous positive pressure ventilation on the non ventilation side, the other groups was ventilation side volume control ventilation+continuous positive pressure ventilation on the non ventilation side; the other groups was ventilation side pressure regulated volume control ventilation+continuous positive pressure ventilation on the non ventilation side.

ELIGIBILITY:
Inclusion Criteria:

Comprehensive examination and analysis of imaging, laboratory examination and other comprehensive examinations, the diagnosis is clear, which is in line with lobe resection surgical indications

Age 18-75 years old, the gender is not limited;

ASA grading Ⅰ ~ III level;

It is expected that the single lung ventilation time is ≥1 hours, and ≤3 hours

Exclusion Criteria:

Emergency surgery;

There is a taboos on the existence of systemic anesthesia;

There is a history of acute chronic upper respiratory infections in the past January;

Previous bronchial asthma, chronic obstructive pulmonary disease, bronchial dilatation, phthisis ,aspergillosis , acute respiratory distress syndrome or history of respiratory failure;

Merge the function of important organs such as heart, liver, and kidney;

There was a history of chest surgery and the history of trauma;

Preoperative lung function test obvious abnormal abnormal abnormalities (1 second of exhalation (FEV1) <60%);

Patients refuse to participate in the clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Clinical Pulmonary Infection Score | Within 15 days after surgery
  The clinical pulmonary infection score index is mainly used to evaluate the severity of pulmonary infection, which involves many factors, including: body temperature, white blood cell count, tracheal secretions, oxygenation, X-ray chest X-ray, and the progress of pulmonary infiltrates. The maximum score is 12 points, and the severity of infection is directly proportional to its score.

CONTACTS AND LOCATIONS:
Overall Officials: Pan Jiamei, Study Director — Staff member of Department of Anesthesiology,Affiliated Hospital of Zunyi Medical University; Zhang Hong, Principal Investigator — Chief physician of Department of Anesthesiology,Affiliated Hospital of Zunyi Medical University
Locations (1):
- Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou, China

IPD SHARING:
Plan to Share IPD: Yes
After the clinical trial , each groups and its clinical pulmonary Infection score were shared with other research teams.
Supporting Information: CSR
Time Frame: Data related to this trial can be shared for a total 6 months after publication.
Access Criteria: Contact the head of the study for approval